CLINICAL TRIAL: NCT01842672
Title: A Pilot Study of Mitoxantrone in Combination With Clofarabine (MITCL) in Children, Adolescents and Young Adults (CAYA) With Refractory/Relapsed Acute Leukemia or High Grade Non-Hodgkin Lymphoma
Brief Title: Mitoxantrone and Clofarabine for Treatment of Recurrent NHL or Acute Leukemia
Acronym: MITCL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC 542; L 10, 819 (Other: New York Medical College Institutional Review Board)
Record Dates: First submitted 2013-04-22; First posted 2013-04-30 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myelogenous Leukemia; Lymphoblastic Lymphoma; Diffuse Large B-cell Lymphoma; Burkitt Lymphoma/Leukemia
Keywords: pediatric non-hodgkins lymphoma; pediatric acute leukemia; clofarabine; mitoxantrone
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma | interventions — Clofarabine; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mitoxantrone/Clofarabine (Experimental): Clofarabine Dose escalation starting 20 mg/m2/d days 1-5 Mitoxantrone 12 mg/m2/d days 3-6. Rituximab in patient with CD20+ disease only 375 mg/m2 day 1, 8, 15. IT Depocyt 35 or 50 mg/dose day 1 per cycle. IT ARA-C in children < 3 years age based dosing.
  Interventions: Drug: Clofarabine; Drug: Mitoxantrone

INTERVENTIONS:
Drug: Clofarabine — Dose Escalation of Clofarabine
  Other Names: Clolar™; Evoltra; NSC# 606,869; IND # 73,789
Drug: Mitoxantrone
  Other Names: Novantrone

SUMMARY:
The combination of mitoxantrone and clofarabine as reinduction therapy will be safe, well tolerated and effective in children, adolescents and young adults with poor risk refractory/relapsed acute leukemia and high grade non-Hodgkin lymphoma (NHL).

ELIGIBILITY:
Inclusion Criteria:

Age ≤30.99 years old

Disease Status (Part A - Safety Phase)

* ALL in 1st, 2nd or 3rd relapse OR primary induction failure.
* AML in 1st ,2nd or 3rd relapse OR primary induction failure.
* T-or B -- Lymphoblastic Lymphoma (T-LBL, B-LBL); Diffuse Large B-cell Lymphoma (DLBCL) or Burkitt Lymphoma/Leukemia in 1st, 2nd or 3rd relapse OR primary induction failure.

5.1.2.2 (Part B - Efficacy Phase)

* ALL in 2nd or 3rd relapse OR primary induction failure.
* AML in 2nd or 3rd relapse OR primary induction failure.
* T-or B -- Lymphoblastic Lymphoma (T-LBL, B-LBL); Diffuse Large B-cell Lymphoma (DLBCL) or Burkitt Lymphoma/Leukemia in 1st, 2nd or 3rd relapse OR primary induction failure.

Adequate renal function defined as:

- Normal Serum creatinine based on age or Creatinine clearance > 60 ml/min or >60 ml/min/1.73 m2 or an equivalent radioisotope glomerular filtration rate (GFR) as determined by the institutional normal range.

Adequate liver function defined as:

* Direct bilirubin < 1.5 upper limit of normal (ULN) for age, and SGOT (AST) or SGPT (ALT) <3 x ULN

Adequate cardiac function defined as:

* Shortening fraction >27% by echocardiogram, or
* Ejection fraction of >50% by radionuclide angiogram or echocardiogram.

Performance Status

* For patients age 1-16 years, Lansky score of ≥60.
* For patients > 16 years, Karnofsky score of ≥60.

Negative urine pregnancy test for females of child bearing age.

Prior Therapy - Patients are eligible if they have been treated with clofarabine, mitoxantrone, or a combination of both in the past. However, the maximal lifetime cumulative previous anthracycline dose should not exceed doxorubicin dose equivalent of 450 mg/m2 (see Table 1). Patients who received more than one anthracycline prior to study entry should have each individual agent cumulative dose converted to doxorubicin equivalent and added together (eg, a patient who received cumulative dose of Daunorubicin at 200 mg/m2 and Mitoxantrone 48 mg/m2 has a total doxorubicin dose equivalent of 358.6 mg/m2 (200 mg/m2 x 0.833 + 48 mg/m2 x 4).

Table 1. Anthracycline Conversion Agent Conversion Factor to Doxorubicin Dose Doxorubicin Multiply total dose x 1 Daunorubicin Multiply total dose x 0.833 Idarubicin Multiply total dose x 5 Mitoxantrone Multiply total dose x 4

Informed Consent

- Patients or the patient's legally authorized guardian must be fully informed about their illness and the investigational nature of this protocol (including foreseeable risks and possible side effects), and must sign an informed consent in accordance with the institutional policies approved by the U.S. Department of Health and Human Services.

Exclusion Criteria:

Patients with prior myeloablative allogeneic stem cell transplantation <3 months prior to proposed enrollment on study and/or ≥Grade II active acute GVHD or extensive chronic GVHD.

Females who are pregnant (positive HCG) or lactating.

Karnofsky <60% or Lansky <60% if less than 16 years of age.

Age >30.99 years of age.

Patients with active CNS disease.

Any patient with uncontrolled infection prior to study entry.

Patients with Down syndrome are excluded.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2013-03; Primary Completion 2021-08 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Determine MTD | 100 days
  2.1 To determine the maximal tolerated dose (MTD) and/or tolerable dose of escalating doses of clofarabine starting from 20mg/m2/day to 40mg/m2/day from Day 1 to Day 5 in combination with mitoxantrone 12mg/m2/day on Day 3-6 as reinduction therapy for children, adolescents and young adults with poor risk refractory/relapsed acute leukemia or high grade NHL.

SECONDARY OUTCOMES:
Response Rate | 1 year
  To determine the overall complete and partial response rate (OR) of the combination of mitoxantrone and clofarabine as reinduction therapy for children, adolescents and young adults with refractory/relapsed acute leukemia or high grade NHL.
Monitor for Minimal Residual Disease | 1 Year
  To determine the percent of minimal residual disease (MRD) in the peripheral blood following reinduction with mitoxantrone and clofarabine reinduction therapy.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - New York Medical College, Valhalla, New York
  - Levine Children's Hospital, Charlotte, North Carolina

REFERENCES:
- [Derived] Hochberg J, Oesterheld J, Gardenswartz A, Flower A, Klejmont L, Basso J, Shi Q, Harrison L, Borowitz MJ, Loken MR, Cairo MS. Mitoxantrone in combination with clofarabine (MITCL) in children, adolescents and young adults with relapsed/refractory acute leukaemia: final results of a phase I/II trial. EClinicalMedicine. 2025 Apr 28;83:103211. doi: 10.1016/j.eclinm.2025.103211. eCollection 2025 May. PMID 40641817